CLINICAL TRIAL: NCT01225328
Title: Participation Restrictions in Young-Middle Adult Rural Breast Cancer Survivors
Brief Title: Participation Restrictions in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: D1032
Record Dates: First submitted 2010-10-19; First posted 2010-10-21 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Telephone-delivered Behavioral Activation/Problem Solving (BA/PS) intervention
  Interventions: Behavioral: Behavioral activation/problem-solving (BA/PS)

INTERVENTIONS:
Behavioral: Behavioral activation/problem-solving (BA/PS) — Six weekly telephone sessions to train participant in BA/PS procedures

SUMMARY:
This project will develop and preliminarily evaluate an intervention to assist young-middle adult rural breast cancer survivors to overcome functional impairments related to their cancer treatment. Younger breast cancer survivors (below age 60) have ongoing family, social and vocational responsibilities and recreational interests and are at increased risk of developing long-term difficulties performing these valued activities (participation restrictions). Rural cancer survivors are medically underserved and due to distance and geographic isolation face significant barriers to accessing traditional rehabilitation services. Alternative rehabilitation approaches are sorely needed for this population. Based on previous research with cancer and other medical populations a working draft of a treatment manual using a telephone-delivered Behavioral Activation and Problem Solving (BA/PS) intervention has been designed. Prior to testing the intervention in a randomized clinical trial, additional work must be completed. The specific aims of this study are to a. refine the BA/PS treatment manual, b. develop and apply treatment integrity measures for the BA/PS manual, c. assess participation restrictions and associated outcomes, d. preliminarily assess the immediate and maintenance effects of BA/PS, and e. examine mediators and moderators of BA/PS effects based on our "Self Regulation" model of functional recovery. 188 young-middle adult breast cancer survivors will be screened for participation restrictions following cancer treatment and 40 survivors with participation restrictions will receive BA/PS delivered by phone. BA/PS participants will be assessed for treatment effectiveness and interviewed regarding their experiences during treatment to provide information for refining the manual. The long-term objective of this line of research is to develop effective and feasible treatments for the medical and psychosocial consequences of cancer and its treatment in medically underserved cancer survivors (e.g., rural populations).

ELIGIBILITY:
Inclusion Criteria:

1. Female breast cancer patient stages I-III.
2. Age 18-59.
3. Completion of definitive breast cancer treatment (i.e., subsequent to loco-regional surgical treatment and completion of adjuvant or neo-adjuvant chemotherapy with or without radiation) within the past 3-6 months.
4. Screen positive for a moderate or worse level of participation restriction (Work and Social Adjustment Scale score > 10) within 6 months following cancer treatment.
5. English speaking.
6. Have a land-based phone or reliable cell phone reception.

Exclusion Criteria:

1. Non-correctable hearing loss.
2. Moderate-severe cognitive impairment indicated by a score < 3 on a 6-item cognitive screener.
3. Medical record documentation of severe mental illness (i.e., schizophrenia or bipolar disorder) or active substance abuse.
4. Medical record documentation of a physical disorder with associated functional impairment (e.g., Parkinson's disease, stroke, congestive heart failure, etc.).

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Feasibility | six weeks
  * of patients evaluated for enrollment / # of patients approached.
  * of patients meeting eligibility criteria / # of patients evaluated.
  * of patients enrolled / # of patients meeting eligibility criteria
  * of patients completing 6 weeks of BA/PS treatment.
  * of patients completing each study assessment point (T1, T2, T3, T4).

SECONDARY OUTCOMES:
Functional status | baseline, six weeks, 12 weeks, 18 weeks
  The Medical Outcomes Short Form-36 (MOS SF-36) consists of eight scales (physical functioning, role limitations - physical, role limitations - emotional, vitality, well being, social functioning, bodily pain, and general health) and two standardized component summary scores (physical and mental). The physical and mental factors account for 80-85% of the variance in the scales. We will use the Physical Component Summary (PCS) Score as the primary outcome measure.
Quality of life | baseline, six weeks, 12 weeks, 18 weeks
  The Functional Assessment of Cancer Therapy-Breast Cancer + Arm Morbidity (FACT-B+4) is a 41-item self-report measure of health-related quality of life specifically designed for breast cancer patients.
Affective symptoms | baseline, six weeks, 12 weeks, 18 weeks
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item self-report measure of depressive and anxiety symptoms specifically designed for medical patients. The HADS contains only the cognitive symptoms of depression and anxiety, thus eliminating the somatic symptoms that are poor indicators of psychiatric distress in the medically ill.

CONTACTS AND LOCATIONS:
Overall Officials: Mark T Hegel, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States